CLINICAL TRIAL: NCT03095222
Title: Exploring the Safety and Efficacy of Low-dose Ketamine Infusions for Pain Control in Acute Burn Injury
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study never screened or enrolled any subjects due to stalled recruitment efforts.
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004424
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2017-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ketamine; Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Daily (Active Comparator): Daily ketamine infusions of 5 hours in length. Duration of participation will last 4 days.
  Interventions: Drug: Ketamine; Drug: Opioids
- Group 2: Continuous (Active Comparator): Continuous ketamine infusions (24 hours/day). Duration of participation will last 4 days.
  Interventions: Drug: Ketamine; Drug: Opioids

INTERVENTIONS:
Drug: Ketamine — To be given as intravenous infusion. Ketamine infusions will be started at 5 mg/hr and can be increased by nursing staff based on patient-reported pain relief up to a maximum hourly rate of 20 mg/hr.
Drug: Opioids — Standard of care for pain management.

SUMMARY:
The purpose of this study is to identify the optimal dosing strategy for low-dose ketamine infusions in adult acute burn injury patients when used with usual pain medications.

DETAILED DESCRIPTION:
This Aim will identify the safest and most optimal dosing strategy for low-dose ketamine infusions. While the hourly rate for low-dose ketamine infusions used for adjunctive analgesia appears to be well-established both in the medical literature and our institutional protocols, there is no information available for this specific population of patients (adult acute burn injury) to know whether the infusions should be utilized for discrete periods of time or should be given continuously. Findings from this study will help provide preliminary data on the optimal dosing strategy of this medication for adjunctive analgesia in this population.

ELIGIBILITY:
Inclusion Criteria:

* Acute burn injury comprising 10-30% of total body surface. Burns severity may include second or third degree burns
* Burn injury must have occurred within 72 hours of enrollment and randomization
* Subjects may be opioid-naïve or opioid non-naïve
* Anticipated stay in the burn unit is greater than 4 days, which is typically the minimum length of stay for patients with this level of burn injury

Exclusion Criteria:

* Burn injury older than 72 hours
* Acute burn injury comprising >30% total body surface
* Patients who are intubated
* Patients who have contraindication to ketamine administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Change in pain severity | Day 4
  Pain severity measured using the 11-point Visual Numerical Scale (VNS). Scores range from 0 to 10. A score of 0 represents no pain. A score of 10 represents the worst pain imaginable. The score will be collected each day. An average of the score will be calculated for all days of the study.

SECONDARY OUTCOMES:
Opioid Analgesic Consumption | Day 4
  All subjects will be on some form of opioid analgesic. All opioid usage will be recorded. For each 24 hour period, the total daily opioid consumption will be calculated and converted to oral morphine equivalents. The outcome will be reported as an average over all days of participation.
Side effects / Adverse effects | Days 1-4
  Any side effects or adverse effects attributed to ketamine infusions will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Nicol, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States